CLINICAL TRIAL: NCT01473420
Title: A Therapeutic-equivalence Study Comparing The Efficacy And Safety Of Subcutaneous Epoetin Hospira And Epoetin Alfa (Amgen) In Patients With Chronic Renal Failure Requiring Hemodialysis And Receiving Epoetin Maintenance Treatment
Brief Title: A Phase 3 Study Comparing the Effects of Subcutaneous Epoetin Hospira and Epoetin Alfa [Epogen] (Amgen) in Patients With Chronic Renal Failure Requiring Hemodialysis and Receiving Epoetin Maintenance Treatment. AiME - Anemia Management With Epoetin
Acronym: AiME - 13
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPOE-10-13; C3461003 (Other: Alias Study Number)
Record Dates: First submitted 2011-11-02; First posted 2011-11-17 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Chronic Renal Failure; Chronic Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epoetin Hospira (Experimental): Epoetin Hospira
  Interventions: Biological: Epoetin Hospira
- Epogen (Amgen) (Active Comparator): Epogen (Amgen)
  Interventions: Biological: Epogen Amgen

INTERVENTIONS:
Biological: Epoetin Hospira — Variable dose
  Arms: Epoetin Hospira
Biological: Epogen Amgen — Variable dose
  Other Names: Epoetin Alfa
  Arms: Epogen (Amgen)

SUMMARY:
The purpose of this study is to demonstrate therapeutic equivalence of subcutaneous (SC) Epoetin Hospira compared to SC Epogen (Amgen), based on maintenance of hemoglobin (Hb) levels and study drug dose requirements in patients treated for anemia associated with chronic renal failure and on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to provide written informed consent after risks and benefits of the study have been explained prior to any study related activities
2. Hemodialysis patients with chronic renal failure and renal anemia currently on stable Epogen (Amgen) dose administered IV or SC, 1 to 3 times per week for whom the following apply:

   * A change in Epogen dosing of no more than 10% from the mean
   * Mean hemoglobin between 9.0 and 11.0 g/dL
   * No more than one hemoglobin result outside of range from 9.0-11.0 g/dL
   * No hemoglobin result more than ±1 g/dL from the mean hemoglobin level
3. Patients on stable, adequate dialysis for at least 12 weeks prior to randomization, defined as no clinically relevant changes of dialysis regimen and/or dialyzer
4. Patients with adequate iron stores, defined as plasma ferritin > 100 μg/L and TSAT >20%, prior to randomization
5. Male or female patients aged 18 to 80 years (both inclusive)
6. If female, patient must be postmenopausal for at least one year prior to randomization, surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or practicing at least one of the following methods of birth control:

   * hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to randomization
   * intrauterine device (IUD)
   * double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream)

If hormonal contraceptives are used, the specific contraceptive must have been used for at least 3 months prior to randomization. If the patient is currently using a hormonal contraceptive, she should also use a barrier method during this study and for at least 30 days following the administration of the patient's last dose

Exclusion Criteria:

1. Maintenance epoetin dosage >600 U/kg per week (1-3 times per week)
2. Treatment with long-acting epoetin analogues such as Aranesp ® within 12 weeks prior to randomization
3. Any of the following within 3 months prior to randomization:

   * Myocardial infarction
   * Stroke (cerebrovascular accident)/cerebrovascular insult (minor stroke) or transient ischemic attack/intracerebral bleeding/cerebral infarction
   * Severe/unstable angina
   * Coronary angioplasty, bypass surgery, or peripheral artery bypass graft
   * Decompensated congestive heart failure (New York Heart Association [NYHA] class IV)
   * Pulmonary embolism
   * Deep vein thrombosis or other thromboembolic event
   * Received live or attenuated vaccination (except flu vaccination)
4. Uncontrolled hypertension within the 4 weeks prior to randomization defined as more than 10% of post-dialysis blood pressures >170 mmHg systolic and/or >110 mmHg diastolic, based on blood pressure readings obtained when the patient's post-dialysis body weight was not more than 0.5 kg above their listed dry weight
5. Known, clinically manifested deficiency of folic acid and/or vitamin B12 (irrespective of whether currently treated or not)
6. A patient with any active, uncontrolled systemic, inflammatory or malignant disease that in the Investigator's opinion may be significant to exclude participation in the study, including but not limited to demyelinating diseases such as multiple sclerosis, microbial, viral or fungal infection or mental disease
7. Contraindication for the test drug or have been previously treated with Epoetin Hospira
8. Relative or absolute iron deficiency prior to randomization into the Maintenance Period
9. Platelet count below 100 x 10^9/L
10. Clinically relevant increase of CRP (>10 mg/dL) for at least 2 weeks
11. Significant drug sensitivity or a significant allergic reaction to any drug, as well as known hypersensitivity or idiosyncratic reaction to epoetin (or its excipients, including albumin) or any other related drugs that in the judgment of the Investigator is exclusionary for the study participation
12. History of any of the following:

    * Detectable anti-rhEPO antibodies
    * Clinically relevant malnutrition
    * Confirmed aluminum intoxication
    * Myelodysplastic syndrome
    * Known bone marrow fibrosis (osteitis fibrosa cystica)
    * Known seizure disorder
    * Liver cirrhosis with clinical evidence of complications (portal hypertension, splenomegaly, ascites)
13. A female patient who is pregnant, lactating or planning a pregnancy during the study
14. History of drug abuse or alcohol abuse within 2 years prior to randomization as determined by the Investigator
15. Current participation or participation in a drug or other investigational research study within 30 days prior to randomization
16. May not be able to comply with the requirements of this clinical study, communicate effectively with study personnel, or is considered by the Investigator, for any reason, to be an unsuitable candidate for the study
17. Donated or lost >475 mL (i.e., 1 pint) blood volume (including plasmapheresis) or had a transfusion of any blood product within 3 months prior to randomization
18. A patient who in the Investigator's opinion, has any clinically significant abnormal laboratory evaluations, including liver function taken at Screening Visit
19. Positive laboratory test for human immunodeficiency virus (HIV) or hepatitis B surface antigen (HBsAg)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2012-01-17 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2014-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (73):
- United States (73):
  - North America Research Institute, Azusa, California
  - National Institute of Clinical Research, Bakersfield, California
  - Long Beach Dialysis Center, Long Beach, California
  - Academic Medical Research Institute, Los Angeles, California
  - Long Beach Dialysis Center, Modesto, California
  - Innovative Dialysis Center of Northridge, LLC, Northridge, California
  - Valley Renal Medical Group, Northridge, California
  - Research Management Inc., Paramount, California
  - Pleasanton Dialysis Center, Pleasanton, California
  - Sunset Dialysis Center, Rancho Cordova, California
  - Capital Nephrology Medical Group, Sacramento, California
  - Chabot Nephrology Medical Group, San Leandro, California
  - San Leandro Dialysis, San Leandro, California
  - Renal Consultants Medical Group, Santa Clarita, California
  - Intercommunity Dialysis Center, Whittier, California
  - American Institute of Research, Whittier, California
  - Whittier Kidney Dialysis Center, Whittier, California
  - Western Nephrology and Metabolic Bone Disease, PC, Arvada, Colorado
  - Kidney Center of Westminster, LLC, Westminster, Colorado
  - Western Nephrology and Metabolic Bone Disease, PC, Westminster, Colorado
  - Pines Clinical Research Inc., Pembroke Pines, Florida
  - Dialysis Clinic, Inc. - Albany, Albany, Georgia
  - Kidney Care Associates, Augusta, Georgia
  - Renal Physicians of Georgia, PC, Dublin, Georgia
  - Neomedica Marquette Park, Chicago, Illinois
  - Research by Design, LLC, Evergreen Park, Illinois
  - Kansas Nephrology Physicians, PA, Wichita, Kansas
  - Research Nurse Specialists, LLC, Lafayette, Louisiana
  - New York Harbor Health Care System, Lafayette, Louisiana
  - Westbank Nephrology Associates, Marrero, Louisiana
  - FMC Opelousas, Opelousas, Louisiana
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - Fresenius Medical Care-Kalamazoo East, Kalamazoo, Michigan
  - Fresenius Medical Care-Kalamazoo, Kalamazoo, Michigan
  - Nephrology Center DBA Paragon Health PC, Kalamazoo, Michigan
  - Fresenius Medical Care-Oshtemo, Kalamazoo, Michigan
  - Fresenius Medical Care-Gull Road, Kalamazoo, Michigan
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Kansas City Renal Center, Kansas City, Missouri
  - Renal Advantage, Inc., Kansas City, Missouri
  - Metro Hypertension and Kidney Center, St Louis, Missouri
  - University of Cincinnati College of Medicine., North Brunswick, New Jersey
  - Nephrology & Hypertension Associates of NJ, Voorhees Township, New Jersey
  - Newtown Dialysis Center, Astoria, New York
  - New York Hospital Medical Center Queens Institutional Review Board, Flushing, New York
  - Parker Jewish Institute for Health Care and Rehabilitation, New Hyde Park, New York
  - New York Harbor Health Care System, New York, New York
  - Wake Nephrology Associates, PA, Raleigh, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Private Practice of Kenneth Lempert, Toledo, Ohio
  - Northwest Physicians Associates, PC, Meadville, Pennsylvania
  - CSRA Renal Services, LLC, Aiken, South Carolina
  - Fresenius Medical Care Midtown JV, Columbia, South Carolina
  - Columbia Nephrology Associates, PA, Columbia, South Carolina
  - Fresenius Medical Care Irmo JV, Irmo, South Carolina
  - South Carolina Nephrology and Hypertension Center, Inc., Orangeburg, South Carolina
  - Knoxville Kidney Center, PLLC, Knoxville, Tennessee
  - Fresenius Medical Care - Austin North Dialysis, Austin, Texas
  - Research Management, Inc., Austin, Texas
  - Research Management, Inc, Austin, Texas
  - Dallas Veterans Affairs Medical Center, Dallas, Texas
  - Grand Prairie Dialysis Center, Grand Prairie, Texas
  - Research Across America, Houston, Texas
  - Westminster Dialysis, Houston, Texas
  - Mission Bend Dialysis, Houston, Texas
  - Southwest Houston Research, Ltd., Houston, Texas
  - East Texas Nephrology Associates, Lufkin, Texas
  - San Antonio Kidney Disease Center, San Antonio, Texas
  - Renal Care Partners of Pentagon City, Arlington, Virginia
  - Clinical Research and Consulting Center, LLC, Fairfax, Virginia
  - Renal Care Partners of Fairfax, Fairfax, Virginia
  - Nephrology Specialists, PC, Mechanicsville, Virginia
  - Western Institutional Review Board, Olympia, Washington

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Wish JB, Rocha MG, Martin NE, Reyes CRD, Fishbane S, Smith MT, Nassar G. Long-term Safety of Epoetin Alfa-epbx for the Treatment of Anemia in ESKD: Pooled Analyses of Randomized and Open-label Studies. Kidney Med. 2019 Aug 28;1(5):271-280. doi: 10.1016/j.xkme.2019.06.009. eCollection 2019 Sep-Oct. PMID 32734207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with chronic renal failure were receiving Epoetin maintenance therapy prior to enrollment and treatment in this study.
Groups:
- Epoetin Hospira: During titration period participants who were on Epogen intravenous (IV) regimen prior to this study, were titrated and optimally stabilized to receive subcutaneous (SC) injection of Epoetin Hospira. Participants who were on Epogen SC regimen prior to this study were continued to receive same as a part of routine clinical practice and did not receive any study treatment during titration period. Dose of study treatment was adjusted to maintain hemoglobin (Hb) level from 9 to 11 gram per deciliter (g/dL). Drug was administered 1 to 3 times per week in titration period (Week 1 to Week 18). During maintenance period participants received SC injection of Epoetin Hospira at optimal dose demonstrated in titration period 1 to 3 times per week up to 16 weeks (Week 19 to Week 34). Participants were followed up to 4 weeks after last dose of study treatment (up to Week 38).
- Epogen: During titration period participants who were on Epogen IV regimen prior to enrollment in this study, were titrated and optimally stabilized to receive SC injection of Epogen. Participants who were on Epogen SC regimen prior to this study were continued to receive same as a part of routine clinical practice and did not receive any study treatment during titration period. Dose was adjusted to maintain the Hb level from 9 to 11 g/dL. Drug was administered 1 to 3 times per week in titration period (Week 1 to Week 18). During maintenance period participants received SC injection of Epogen at the optimal dose demonstrated in the titration period 1 to 3 times per week up to 16 weeks (Week 19 to Week 34). Participants were followed up to 4 weeks after last dose of study treatment (up to Week 38).
Period: Titration Period (18 Weeks)
Arm/Group | Epoetin Hospira | Epogen
Started | 160 | 160
Treated | 80 | 86
Completed | 124 | 122
Not Completed | 36 | 38
Not completed — Adverse Event | 4 | 6
Not completed — Did not meet criteria | 32 | 32
Period: Maintenance Period (16 Weeks)
Arm/Group | Epoetin Hospira | Epogen
Started | 124 | 122
Completed | 106 | 105
Not Completed | 18 | 17
Not completed — Adverse Event | 3 | 2
Not completed — Physician Decision | 1 | 2
Not completed — Did not meet criteria | 0 | 2
Not completed — Kidney transplant | 3 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Site closure | 3 | 1
Not completed — Started Peritoneal Dialysis | 1 | 0
Not completed — Long term hospitalization | 0 | 1
Not completed — Sponsor's Decision | 1 | 0
Not completed — Elevated Hemoglobin | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants who were enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Epoetin Hospira | Epogen | Total
Number analyzed (Participants) | 160 | 160 | 320
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 109 | 117 | 226
  >=65 years | 51 | 43 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 84 | 161
  Male | 83 | 76 | 159

OUTCOME MEASURES:

1. Primary Outcome: Mean Weekly Hemoglobin Level From Week 30 to Week 34: Maintenance Period
Time Frame: Week 30 up to Week 34
Population: This outcome measure was planned not to be analyzed in titration period. Intent-to-treat (ITT) population included all participants who were randomized into the maintenance period.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Epoetin Hospira: Maintenance Period: During maintenance period participants received SC injection of Epoetin Hospira at the optimal dose demonstrated in the titration period. Dose was adjusted to maintain the Hb level from 9 to 11 g/dL. Drug was administered 1 to 3 times per week up to 16 weeks (Week 19 to Week 34). Participants were followed up to 4 weeks after last dose of study treatment (up to Week 38).
- Epogen: Maintenance Period: During maintenance period participants received SC injection of Epogen at the optimal dose demonstrated in the titration period. Dose was adjusted to maintain the Hb level from 9 to 11 g/dL. Drug was administered 1 to 3 times per week up to 16 weeks (Week 19 to Week 34). Participants were followed up to 4 weeks after last dose of study treatment (up to Week 38).
Arm/Group | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 124 | 122
g/dL | 10.17 (0.821) | 10.11 (0.838)
Statistical Analysis 1: Comparison: Epoetin Hospira: Maintenance Period vs Epogen: Maintenance Period; Least square (LS) mean and 95 percent confidence interval (CI) derived from an analysis of covariance (ANCOVA) model with fixed effect of treatment; Test type: Non-Inferiority or Equivalence — An equivalence margin of +/- 0.5 was considered relevant to demonstrate the equivalence of the two products; LS Mean Difference = 0.04, 95% CI 2-sided [-0.17 to 0.24], Standard Error of Mean 0.104

2. Primary Outcome: Mean Weekly Dosage of Study Medication From Week 30 to Week 34: Maintenance Period
Time Frame: Week 30 up to Week 34
Population: This outcome measure was planned not to be analyzed in titration period. ITT population included all participants who were randomized into the maintenance period.
Measure: Mean (Standard Deviation); unit: unit per kilogram per week (U/kg/week)
Arm/Group | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 124 | 122
unit per kilogram per week (U/kg/week) | 82.07 (95.517) | 79.14 (82.264)
Statistical Analysis 1: Comparison: Epoetin Hospira: Maintenance Period vs Epogen: Maintenance Period; LS mean and 95 percent CI derived from an ANCOVA model with fixed effect of treatment; Test type: Non-Inferiority or Equivalence — An equivalence margin of +/- 0.5 was considered relevant to demonstrate the equivalence of the two products; LS Mean Difference = -2.34, 95% CI 2-sided [-14.51 to 9.82], Standard Error of Mean 6.175

3. Secondary Outcome: Mean Weekly Hemoglobin Level From Week 19 to Week 34: Maintenance Period
Time Frame: Week 19 up to Week 34
Population: This outcome measure was planned not to be analyzed in titration period. ITT population included all participants who were randomized into the maintenance period. Here, "Number of Participants Analyzed" (N) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 124 | 121
g/dL | 10.20 (0.625) | 10.22 (0.665)
Statistical Analysis 1: Comparison: Epoetin Hospira: Maintenance Period vs Epogen: Maintenance Period; Test type: Superiority or Other; p = 0.8338, Two-sample t-test

4. Secondary Outcome: Mean Weekly Dosage of Study Medication From Week 19 to Week 34: Maintenance Period
Time Frame: Week 19 up to Week 34
Population: This outcome measure was planned not to be analyzed in titration period. ITT population included all participants who were randomized into the maintenance period. Here, "N" signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: U/kg/week
Arm/Group | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 123 | 121
U/kg/week | 81.93 (93.824) | 75.08 (72.174)
Statistical Analysis 1: Comparison: Epoetin Hospira: Maintenance Period vs Epogen: Maintenance Period; Test type: Superiority or Other; p = 0.6895, Wilcoxon Rank Sum test; P-value was calculated from a Wilcoxon Rank Sum test and t-approximation was used

5. Secondary Outcome: Total Dose of Study Medication Administered: Maintenance Period
Description: In this outcome measure mean of total dose of study medication administered in maintenance period was reported.
Time Frame: Week 19 up to Week 34
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units of study medication
Arm/Group | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 123 | 121
units of study medication | 102003.2 (135560.52) | 86478.5 (83351.03)
Statistical Analysis 1: Comparison: Epoetin Hospira: Maintenance Period vs Epogen: Maintenance Period; Test type: Superiority or Other; p = 0.9177, Wilcoxon Rank Sum test; P-value was calculated from a Wilcoxon Rank Sum test and t-approximation was used

6. Secondary Outcome: Percentage of Participants With Mean Weekly Hemoglobin Level Within the Target Range: Maintenance Period
Description: Percentage of participants who had hemoglobin level within the target range of 9 to 11 g/dL for the specified weeks were reported.
Time Frame: Week 26, 34
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 124 | 122
percentage of participants
  Week 26 | 73.5 | 60.9
  Week 34 | 79.8 | 74.0

7. Secondary Outcome: Percentage of Participants Who Required Permanent Dose Changes: Maintenance Period
Time Frame: Week 19 up to Week 34
Population: This outcome measure was planned not to be analyzed in titration period. Per protocol population included all participants who were randomized into the maintenance period and who did not have major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 86 | 92
percentage of participants | 30.2 | 25.0

8. Secondary Outcome: Percentage of Participants Who Required Temporary Dose Changes: Maintenance Period
Time Frame: Week 19 up to Week 34
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 86 | 92
percentage of participants | 55.8 | 62.0

9. Secondary Outcome: Percentage of Participants With Any Transient Change of Hemoglobin Level Greater Than (>) 1.0 Gram Per Deciliter (g/dL): Maintenance Period
Time Frame: Week 19 up to Week 34
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 86 | 92
percentage of participants | 29.1 | 52.2

10. Secondary Outcome: Percentage of Participants With Mean Weekly Hemoglobin Level Outside the Target Range: Maintenance Period
Description: Percentage of participants who had hemoglobin level outside the target range of 9 to 11 g/dL for the specified weeks were reported.
Time Frame: Week 26, 34
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 124 | 122
percentage of participants
  Week 26 | 13.5 | 19.3
  Week 34 | 10.1 | 13.0

11. Secondary Outcome: Percentage of Participants Who Qualified as Optimally Titrated and Stable: Titration Period
Time Frame: Week 1 up to Week 18
Population: This outcome measure was planned not to be analyzed in maintenance period. Safety analysis population for titration period included all participants who received at least 1 dose of study treatment in titration period.
Measure: Number; unit: percentage of participants
Groups:
- Epoetin Hospira: Titration Period: During titration period participants who were on Epogen IV regimen prior to this study, were titrated and optimally stabilized to receive SC injection of Epoetin Hospira. Participants who were on Epogen SC regimen prior to this study were continued to receive same as a part of routine clinical practice and did not receive any study treatment during titration period. Dose of study treatment was adjusted to maintain Hb level from 9 to 11 g/dL. Drug was administered 1 to 3 times per week in titration period (Week 1 to Week 18).
- Epogen: Titration Period: During titration period participants who were on Epogen IV regimen prior to enrollment in this study, were titrated and optimally stabilized to receive SC injection of Epogen. Participants who were on Epogen SC regimen prior to this study were continued to receive same as a part of routine clinical practice and did not receive any study treatment during titration period. Dose was adjusted to maintain the Hb level from 9 to 11 g/dL. Drug was administered 1 to 3 times per week in titration period (Week 1 to Week 18).
Arm/Group | Epoetin Hospira: Titration Period | Epogen: Titration Period
Number analyzed (Participants) | 80 | 86
percentage of participants | 47.5 | 47.7

12. Secondary Outcome: Percentage of Participants Who Received Blood Transfusions: Maintenance Period
Time Frame: Week 19 up to Week 34
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 124 | 122
percentage of participants | 4.0 | 4.1

13. Secondary Outcome: Number of Participants With Change in Mean Dose of Study Medication Based on Hemoglobin Level: Maintenance Period
Description: In this outcome measure number of participants with change (increase and decrease) in mean dose of Epoetin Hospira and Epogen were categorized and reported according to their mean hemoglobin levels. Hemoglobin levels were divided in following classes: >11.0 g/dL, from 9.0 to 11.0 g/dL and <9.0 g/dL
Time Frame: Week 19 up to Week 34
Population: This outcome measure was planned not to be analyzed in titration period. ITT population included all participants who were randomized into the maintenance period. Here, "N" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 123 | 121
Participants
  Dose Decrease: Hb <9.0 g/dL | 9 | 10
  Dose Decrease: Hb (9.0 to 11.0 g/dL) | 20 | 14
  Dose Decrease: Hb >11.0 g/dL | 35 | 40
  Dose Increase: Hb <9.0 g/dL | 24 | 23
  Dose Increase: Hb (9.0 to 11.0 g/dL) | 11 | 3
  Dose Increase: Hb >11.0 g/dL | 7 | 13

14. Secondary Outcome: Percentage of Participants With Any Transient Change of Hemoglobin Level Greater Than (>) 2.0 Gram Per Deciliter (g/dL) in Hemoglobin Level: Maintenance Period
Time Frame: Week 19 up to Week 34
Population: This outcome measure was planned not to be analyzed in titration period. Safety analysis population for maintenance period included all participants who received at least 1 dose of study treatment in maintenance period.
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 122 | 122
percentage of participants | 6.6 | 10.7

15. Other Pre Specified Outcome: Percentage of Participants With Hemoglobin Level Less Than (<) 8.0 Gram Per Deciliter (g/dL): Maintenance Period
Time Frame: Week 19 up to Week 34
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 122 | 122
percentage of participants | 4.1 | 9.0

16. Other Pre Specified Outcome: Percentage of Participants With Hemoglobin Level Greater Than (>) 12.0 Gram Per Deciliter (g/dL): Maintenance Period
Time Frame: Week 19 up to Week 34
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 122 | 122
percentage of participants | 9.8 | 19.7

17. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Titration Period: Week 1 up to Week 18 and Maintenance Period: Week 19 up to Week 38
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira: Titration Period | Epogen: Titration Period | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 80 | 86 | 122 | 122
Participants
  AEs | 45 | 54 | 85 | 86
  SAEs | 12 | 22 | 23 | 33

18. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events by Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. An AE was assessed according to severity; mild (AE was transient and easily tolerated by the participant), moderate (caused problem that did not interfere significantly with usual activities) and severe (caused problem that interferes significantly with usual activities and might be incapacitating or life-threatening).
Time Frame: Titration Period: Week 1 up to Week 18 and Maintenance Period: Week 19 up to Week 38
Population: Safety population included all participants who received at least 1 dose of study treatment. Here, "N" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira: Titration Period | Epogen: Titration Period | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 45 | 54 | 85 | 86
Participants
  Mild | 21 | 23 | 42 | 41
  Moderate | 15 | 16 | 24 | 27
  Severe | 9 | 15 | 19 | 18

19. Other Pre Specified Outcome: Number of Participants With Treatment Related Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug.
Time Frame: Titration Period: Week 1 up to Week 18 and Maintenance Period: Week 19 up to Week 38
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira: Titration Period | Epogen: Titration Period | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 45 | 54 | 85 | 86
Participants | 1 | 4 | 7 | 11

20. Other Pre Specified Outcome: Number of Participants That Discontinued Treatment Due to a Treatment Emergent Adverse Event
Description: In this outcome measure number of participants discontinued from study drug (Epoetin Hospira, Epogen) due to any AE were reported.
Time Frame: Titration Period: Week 1 up to Week 18 and Maintenance Period: Week 19 up to Week 38
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira: Titration Period | Epogen: Titration Period | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 45 | 54 | 85 | 86
Participants | 4 | 6 | 4 | 4

21. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Parameters
Description: Laboratory parameters: Hematology (hematocrit, hemoglobin, red blood cell count, reticulocytes, white blood cell count, neutrophils, bands, lymphocytes, monocytes, basophils, eosinophils, platelet count, mean corpuscular volume); coagulation panel (prothrombin time, international normalized ratio, activated partial thromboplastin time); clinical chemistry (blood urea nitrogen, creatinine, alanine aminotransferase, aspartate aminotransferase, total bilirubin, gamma-glutamyl transpeptidase, alkaline phosphatase, sodium, potassium, calcium, magnesium, phosphorus, uric acid, total protein, glucose, albumin, C-reactive protein, plasma ferritin, transferrin saturation). Participants with clinically significant change from baseline in laboratory parameters were as determined by the investigator.
Time Frame: Titration Period: Baseline (Pre-dose on Week 1) up to Week 18 and Maintenance Period: Baseline (Pre-dose on Week 19) up to Week 38
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira: Titration Period | Epogen: Titration Period | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 80 | 86 | 122 | 122
Participants | 0 | 0 | 0 | 0

22. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital sign parameters: temperature (oral, tympanic, or other), blood pressure (diastolic and systolic), heart rate (in a seated position) and dry weight (post-dialysis). Participants with clinically significant change from baseline in vital signs were as determined by the investigator.
Time Frame: as for outcome 21
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira: Titration Period | Epogen: Titration Period | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 80 | 86 | 122 | 122
Participants | 0 | 0 | 0 | 0

23. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG)
Description: ECG parameters: PR interval, QRS complex, QT interval and QTC interval. Participants with clinically significant change from baseline in ECG were as determined by the investigator.
Time Frame: as for outcome 21
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira: Titration Period | Epogen: Titration Period | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 80 | 86 | 122 | 122
Participants | 0 | 0 | 0 | 0

24. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examination
Description: Physical examination included examination of the following: skin, eyes, ears, throat, cardiac, respiratory, gastrointestinal, genitourinary and musculoskeletal systems. Participants with clinically significant change from baseline in physical examination were as determined by the investigator.
Time Frame: as for outcome 21
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira: Titration Period | Epogen: Titration Period | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 80 | 86 | 122 | 122
Participants | 0 | 0 | 0 | 0

25. Other Pre Specified Outcome: Percentage of Participants With Anti-Recombinant Human Erythropoietin (Anti-rhEPO) Antibodies
Description: Percentage of participants with presence of anti-rhEPO antibodies were reported in this outcome measure. Radioimmunoprecipitation assay method was used to determine the presence of anti-rhEPO antibodies.
Time Frame: Titration Period: Week 1 up to Week 18 and Maintenance Period: Week 19 up to Week 38
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira: Titration Period | Epogen: Titration Period | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 34 | 36 | 104 | 108
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

26. Other Pre Specified Outcome: Percentage of Participants With General Tolerability
Description: General tolerability was classified as: 1) excellent tolerability = no reaction, 2) good tolerability = minimal reaction, 3) mild intolerability = reaction above that normally observed with any kind of subcutaneous product, 4) moderate intolerability = marked reaction, but no need for discontinuation of treatment and 5) severe intolerability = treatment discontinued due to intolerability.
Time Frame: Titration Period: Week 1 up to Week 18 and Maintenance Period: Week 19 up to Week 38
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira: Titration Period | Epogen: Titration Period | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 80 | 84 | 119 | 121
percentage of participants
  Excellent Tolerability | 68.8 | 67.4 | 63.9 | 50.8
  Good Tolerability | 28.8 | 25.6 | 27.0 | 27.9
  Mild Intolerability | 2.5 | 2.3 | 4.9 | 16.4
  Moderate Intolerability | 0.0 | 2.3 | 0.0 | 2.5
  Severe Intolerability | 0.0 | 0.0 | 1.6 | 1.6

27. Other Pre Specified Outcome: Percentage of Participants With Local Tolerability
Description: Local tolerability was classified as: 1) excellent tolerability = no reaction at site of injection, 2) good tolerability = minimal reaction at site of injection normally observed with any kind of subcutaneous product, 3) mild intolerability = reaction at site of injection above that normally observed with any kind of subcutaneous product, 4) moderate intolerability = marked reaction, but no need for discontinuation of treatment and 5) severe intolerability = treatment discontinued due to intolerability.
Time Frame: Titration Period: Week 1 up to Week 18 and Maintenance Period: Week 19 up to Week 38
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira: Titration Period | Epogen: Titration Period | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Number analyzed (Participants) | 80 | 84 | 119 | 121
percentage of participants
  Excellent Tolerability | 70.0 | 66.3 | 67.2 | 54.1
  Good Tolerability | 25.0 | 25.6 | 24.6 | 30.3
  Mild Intolerability | 3.8 | 5.8 | 4.1 | 9.0
  Moderate Intolerability | 1.3 | 1.2 | 1.6 | 3.3
  Severe Intolerability | 0.0 | 0.0 | 0.0 | 2.5

ADVERSE EVENTS:
Description: Same event may appear as both AE and SAE. What is presented are distinct events. An event may be categorized as serious in 1 participant and as non serious in another participant, or 1 participant may have experienced both a serious and non serious event during the study. Safety population.
Arm/Group | Epoetin Hospira: Titration Period | Epogen: Titration Period | Epoetin Hospira: Maintenance Period | Epogen: Maintenance Period
Serious Adverse Events (participants affected / at risk) | 12/80 | 22/86 | 23/122 | 33/122
Other Adverse Events (participants affected / at risk) | 16/80 | 10/86 | 27/122 | 24/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Epoetin Hospira: Titration Period (N=80) | Epogen: Titration Period (N=86) | Epoetin Hospira: Maintenance Period (N=122) | Epogen: Maintenance Period (N=122)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Angina Unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 1 | 2
Cardiac Arrest (Cardiac disorders) | 1 | 1 | 2 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac Perforation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 0 | 0 | 2
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 1 | 2 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 2 | 0
Gangrene (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 3 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 1 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1
Arteriovenous Fistula Occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Graft Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vascular Graft Thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood Culture Positive (Investigations) | 0 | 0 | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Carcinoid Tumour Of The Stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cervical Cord Compression (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Hepatic Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Mental Impairment (Nervous system disorders) | 0 | 0 | 1 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal Cyst Haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Aortic Stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Jugular Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Vena Cava Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 2 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Gastrointestinal Angiodysplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Colon Gangrene (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Graft Infection (Infections and infestations) | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Necrotising Fasciitis (Infections and infestations) | 1 | 0 | 0 | 0
Oesophageal Candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 2 | 0 | 0
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Graft Thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb Traumatic Amputation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/40 | 1/40 | 0/59 | 0/67 — This event was gender specific.
Vulval Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/40 | 0/40 | 0/59 | 0/67 — This event was gender specific.
Vulval Cancer Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/40 | 1/40 | 0/59 | 0/67 — This event was gender specific.
Metabolic Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0/40 | 1/40 | 0/59 | 0/67 — This event was gender specific.
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Aneurysm Ruptured (Vascular disorders) | 0 | 1 | 0 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Hospira: Titration Period (N=80) | Epogen: Titration Period (N=86) | Epoetin Hospira: Maintenance Period (N=122) | Epogen: Maintenance Period (N=122)
Headache (Nervous system disorders) | 4 | 4 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 0 | 3 | 8
Nausea (Gastrointestinal disorders) | 0 | 0 | 10 | 8
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 8 | 3
Injection Site Pain (General disorders) | 0 | 0 | 3 | 8
Pyrexia (General disorders) | 0 | 0 | 8 | 3
Procedural Hypotension (Injury, poisoning and procedural complications) | 5 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 0
Eosinophil Count Increased (Investigations) | 4 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.